CLINICAL TRIAL: NCT00473720
Title: Phase I Dose Finding Study of the Orally Bioavailable Platinum Analog Satraplatin in Combination With Abraxane (Paclitaxel Protein-bound Particles) in Advanced Cancers
Brief Title: Phase I Study of the Combination of Satraplatin and Abraxane in Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Agennix (Industry)
Responsible Party: Principal Investigator, Hari Deshpande, Assistant Professor of Medicine, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0606001535
Record Dates: First submitted 2007-05-11; First posted 2007-05-15 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Cancers
MeSH Terms: interventions — satraplatin; Platinum; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- satraplatin abraxane (Experimental): Satraplatin and abraxane will be given in escalating cohorts on a 3 + 3 design from satraplatin 40mg/m2 and abraxane 80mg/m2
  Interventions: Drug: Satraplatin; Drug: Abraxane

INTERVENTIONS:
Drug: Satraplatin — Dose escalation of 40, 60 and 80 mg/m²/day on days 1-5
  Other Names: platinum analog
Drug: Abraxane — Dose escalation of 80 and 100 mg/mm²/day on days 1,8,15,22 every 28 days
  Other Names: Paclitaxel protein-bound particles

SUMMARY:
This is a phase I dose escalating study of oral satraplatin in combination with Abraxane administered weekly for three out of every four weeks in patients with advanced solid cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed advanced solid tumors.
* The patients must be refractory to standard therapy or have a tumor for which no therapy with clinical benefit exists.
* Patients should have evidence of disease progression if they received a prior therapy. This includes development of new lesions or an increase in preexisting lesions on bone scintigraphy, CT, MRI or by physical examination. Patients in whom the sole criterion for progression is an increase in a biochemical marker, e.g., carcinoembryonic antigen (CEA), or an increase in symptoms, are not eligible, with the exception of the biochemical marker PSA (prostate specific antigen).
* No radiotherapy, treatment with cytotoxic agents, or treatment with biologic agents within the 4 weeks prior to beginning treatment on this study (6 weeks for mitomycin or nitrosoureas). Patients must have fully recovered from the acute toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤ grade 1 are eligible.
* All non-prostate cancer patients need to be at least 2 weeks off any hormonal therapy. Prostate cancer patients need to be maintained with castrate levels of testosterone and at least 2 weeks off any non steroidal anti-androgen, diethylstilbestrol, or ketoconazole.
* At least 2 weeks must have elapsed from any prior surgery .
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%).
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

Hemoglobin ≥ 9 g/dL leukocytes ≥3,000/mcL absolute neutrophil count ≥1,500/mcL platelets ≥100,000/mcL total bilirubin within normal institutional limits AST(SGOT)/ALT(SGPT) ≤2.5 x institutional upper limit of normal creatinine within 1.5 x ULN OR creatinine clearance ≥50 mL/min/1.73 m² for patients with creatinine levels above institutional normal.

* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Pregnant and nursing patients are excluded because the effects of the combination of Abraxane and Satraplatin on a fetus or nursing child are unknown. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Sexually active men must also use appropriate contraception method and should not father a child while receiving therapy during this study.
* Must be able to understand and sign a written informed consent document.

Exclusion Criteria:

* Patients who are less than 4 weeks from chemotherapy or radiotherapy, or have not recovered from any adverse events
* Patients receiving any other investigational agents.
* Patients with known active brain metastases. Patients with treated brain metastases are eligible if they have received radiation to the brain or surgery, more than 4 weeks prior to enrollment onto this study, and do not have progression of their central nervous system disease radiologically or clinically. Such patients should be off steroids for a minimum of two weeks prior to the first dose on study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
* Peripheral neuropathy ≥ Grade 2
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the investigational agents may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated.
* HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy and the potential pharmacokinetic interaction between antiretroviral therapy and the investigational agents.
* Concomitant use of certain medications that inhibit the liver microsomal enzyme CYP3A4 and CYP2CA8/9 may result in increased levels of Satraplatin and/or Abraxane. This increase may be clinically relevant because toxicities are related to dose and exposure. Therefore, all herbal and alternative medications should be discontinued while on study, these include: Hydrastis canadensis (goldenseal), Uncaria tomentosa (cat's claw), Echinacea angustifolia roots, trifolium pratense (wild cherry), matricaria chamomila (chamomile), and Glycyrrhiza glabra (licorice), dillapiol, and naringenim. No concomitant use of the following drugs is allowed: cyclosporine, diltiazem, ketoconazole, rifampin, fluconazole, delavirdine, nicardipine, pioglitazone, and sulfonamides, St Johns Wort. Consumption of grapefruit juice is prohibited during the study. Patients will be asked as to which medicines (traditional or herbal) they are taking at every study visit. If possible, these medications and/or all herbal medicines should not be restarted until 72 hours after the last drug dose on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To determine a safe dose of oral Satraplatin to be administered for 5 consecutive days every week in combination with a 30 minute infusion of Abraxane administered weekly for 3 weeks out of 4 weeks. | Upon completion of dose escalation and determination of MTD

SECONDARY OUTCOMES:
To determine the toxicity profile of Satraplatin combined with Abraxane | Upon completion of study
To determine the anti-tumor effect of the combination of Satraplatin and Abraxane | Upon completion of study
To determine if the administration of Satraplatin alters the pharmacokinetic profile of weekly Abraxane | Upon completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Hari Deshpande, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, Comprehensive Cancer Center, New Haven, Connecticut, United States